CLINICAL TRIAL: NCT06050642
Title: PRO-DIAB-1: Study of the Impact of PROximity Support for Patients With Type 1 DIABetes Treated With an Insulin Pump or Closed Loop.
Brief Title: Study of the Impact of PROximity Support for Patients With Type 1 DIABetes Treated With an Insulin Pump or Closed Loop.
Acronym: PRO-DIAB-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: timkl (Industry)
Collaborators: Sanoia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO-DIAB-1; 2023-A00891-44 (Other: ANSM)
Record Dates: First submitted 2023-09-01; First posted 2023-09-22 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: type 1 diabetes; diabetes distress; insulin pump; insuline closed-loop; home support provider; quality of life; disease burden; treatment satisfaction; Time in Range; Patient-Physician interactions; Pharmacist
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: pragmatic, randomized, prospective, multisite (national), real-life study comparing home support service models
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (Standard Care) (No Intervention): these patients will continue with their current home support provider's standard care
- Interventional arm (Enhanced Care) (Experimental): these patients will be prescribed the enhanced care model to replace the standard care provided by their current home support provider. Patients are informed that they can return to standard care at the end of the study period (1 year), or at any time if they wish to leave the study.
  Interventions: Other: enhanced care model provided by Timkl, a home support provider

INTERVENTIONS:
Other: enhanced care model provided by Timkl, a home support provider — A new type of care provided by timkl, a home support provider, involving nurses and the dispensing pharmacist. This approach combines the current tasks of the service provider's nurses with closer monitoring by the pharmacist, thanks to more frequent contacts and a holistic view of the patient.
  Arms: Interventional arm (Enhanced Care)

SUMMARY:
Amidst medical innovations, many Type 1 diabetes patients using advanced therapy show improved control but still suffer from diabetes-related distress. To tackle this, the investigators propose an "enhanced care" model involving healthcare providers and pharmacists. The study compares standard and enhanced care for Type 1 adults, focusing on the pharmacist's role.

The main question it aims to answer is : In patients with type 1 diabetes treated with pump or closed-loop therapy, does the improved enhanced care versus conventional layout improve diabetes-related distress at 12 months?

Participants will complete a monthly online questionnaire to assess their diabetes-related distress as well as their frequency of use of standard and enhanced care as well as the associated patient satisfaction.

DETAILED DESCRIPTION:
Amidst accelerating innovations in care and limited medical time, many patients with Type 1 diabetes treated by pump or closed-loop therapy appear to have improved glycaemic control, but still experience significant diabetes-related distress.

The investigators therefore propose that a new form of patient care service provided by a health service provider and the patient's pharmacist, as part of the new type of care called "enhanced care", could contribute to overcoming this challenge.

This study compares two different care services provided to adult patients with Type 1 diabetes (PwT1D) treated with an insulin pump or a closed-loop system, known as standard care and enhanced care, the main difference between which lies in the pharmacist's involvement in the enhanced care model.

The originality of this project lies in several points:

* Firstly, it involves evaluating a new care model called enhanced care, which has the original feature of including the involvement of the patient's dispensing pharmacist.
* The role of home support providers in the psychological aspects of diabetes is poorly documented in the scientific literature.

Diabetes-related distress is a well-known complication, but means of prevention remain inadequate. This study integrates live collection of patient data, by the patient. Patient experience is an innovative approach that plays an increasingly important role in the evaluation of new management approaches.

* In addition to patient data, this study integrates data from pharmacists and physicians. These data will be used to compare the points of view of healthcare professionals and patients, in order to gain a precise idea of the service provided by the enhanced care. In itself, this comparison could contribute to identifying and understanding the difference in the points of view of healthcare professionals and patients.
* While there is a wealth of literature demonstrating the value of pharmacist involvement in the care of Type 2 diabetic patients, such information is lacking for Type 1 diabetes. This study, aimed at investigating the impact of the pharmacist, specifically on the distress of patients undergoing highly technical treatment, is therefore original.
* Finally, the design of this pragmatic, randomized study enables real-life practices to be analyzed, while maintaining the highest possible level of evidence.

ELIGIBILITY:
Inclusion Criteria:

* Be an adult (age ≥ 18 years)
* Have Type 1 diabetes
* Have been on closed-loop or insulin pump therapy for ≥ 6 months
* Be in moderate or high diabetes-related distress defined as a DDS2 score ≥ 6
* Be able to understand and complete questionnaires in French
* Be affiliated to the general French Social Security system
* Have an e-mail address
* Have a cell phone number

Non-inclusion criteria:

* Be deprived of liberty, under guardianship or curatorship
* Not have Internet access or a cell phone
* Have benefited or are already benefiting from the Enhanced Care program
* Participating in an interventional study on a medical device for diabetes (pump, sensors, etc.)
* Patients who are not regularly monitored in the investigating center proposing to include them, or who are likely to change centers or move to a different living area (pharmacy) within a year of inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in the 7-question Type-1 Diabetes Distress Score (T1-DDS-7) [Comparison: Enhanced Care vs Standard Care] | Baseline visit (Month 0) to Final visit (Month 12)
  Compare patient-reported levels of diabetes-related distress at 12 months. Higher T1-DDS-7 scores indicate higher levels of diabetes-related distress.

SECONDARY OUTCOMES:
A.1 Change in the 7-question Type-1 Diabetes Distress Score (T1-DDS-7) [Comparison: Enhanced Care vs Standard Care] | Baseline (Month 0) to Month 6
  Compare patient-reported levels of diabetes-related distress at 6 months. Higher T1-DDS-7 scores indicate higher levels of diabetes-related distress.
A.2 Change in the sub-scores of the 7-question Type-1 Diabetes Distress Score (T1-DDS-7) [Comparison: Enhanced Care vs Standard Care] | Baseline (Month 0) to Month 12
  Compare the dimensions of patient-reported levels of diabetes-related distress individually at 12 months.
  Each question of the T1-DDS-7 reports a different dimension of diabetes-related distress.
  Higher sub-scores indicate higher levels of diabetes-related distress in their respective dimensions.
A.3a Evolution of the 7-question Type-1 Diabetes Distress Score (T1-DDS-7) [Comparison: Enhanced Care vs Standard Care] | quarterly between Baseline (Month 0) and Month 12
  Time-series analysis of the evolution of T1-DDS-7 scores over the course of the 12-month observation period. T1-DDS-7 is assessed quarterly. Higher T1-DDS-7 scores indicate higher levels of diabetes-related distress.
A.3b Evolution of the 2-question Diabetes Distress Score (DDS2) [Comparison: Enhanced Care vs Standard Care] | 8 times between Baseline (Month 0) and Month 12
  Time-series analysis of the evolution of DDS2 scores over the course of the 12-month observation period. Higher scores indicate higher levels of diabetes-related distress. DDS2 is every month during which the T1-DDS-7 is not.
  This time series will be used to complete the time-series of T1-DDS-7 scores.
B.1a Patient overall satisfaction with services provided by the home support provider | monthly between Baseline (Month 0) and Month 12
  Overall satisfaction is assessed using a Visual Analog Score ranging from 0 to 10, with higher values indicating higher satisfaction.
B.1b Frequency of patients' interactions with the home support provider | monthly between Baseline (Month 0) and Month 12
  Number of contacts with a representative of the home support provider during the previous month.
  Representatives include : nurses, psychologists, and pharmacists (intervention group only).
B.1c Satisfaction with specific aspects of the services provided by the home support provider | monthly between Baseline (Month 0) and Month 12
  The following aspects of services provided were each assessed using a 5-point Likert scale, ranging from "completely satisfied" to "completely dissatisfied":
  * Were the interactions appropriately personalized for the patient?
  * Were the interactions of adequate quality?
  * Did the patient feel they could trust the representative?
  * Were the interactions of an appropriate length?
  * Was the location of the interactions satisfactory?
  * Was the organization of the interactions satisfactory?
  * Was the number of the interactions satisfactory? The above Likert values may be averaged to provide an overall satisfaction score.
B.2a (Intervention group only) Number of pharmacy visits | monthly between Baseline (Month 0) and Month 12
  To describe the actual intervention during the study, each visit will be reported in the online SanoWeb system.
  The number of pharmacy visits per patient will be counted using SanoWeb data.
B.2b (Intervention group only) Duration of pharmacy visits | monthly between Baseline (Month 0) and Month 12
  The duration of pharmacy visits will be evaluated using SanoWeb data.
B.2c (Intervention group only) Description of clinical or non-clinical events impacting diabetes | monthly between Baseline (Month 0) and Month 12
  During pharmacy visits, patients will have the opportunity to report clinical and non-clinical events. These events are recorded in the SanoWeb system.
B.3a Patients' Perceived Effectiveness of Patient-Physician Interactions (PEPPI questionnaire) | at Month 6 and at Month 12
  The PEPPI questionnaire will be used to assess patients' perceived effectiveness of their interactions with their diabetes specialist. Higher scores indicate better perceived efficacy.
B.3b Patient Assessment of Chronic Illness Care (PACIC questionnaire) | at Baseline (Month 0) and at Month 12
  The PACIC questionnaire will be used to obtain patients' assessment of overall management. Higher scores indicate a better assessment of care.
B.3c Patient assessment of information flow and transparency | at Month 6 and at Month 12
  5-point Likert scale, ranging from "completely satisfied" to "completely dissatisfied"
B.3d Patient assessment of how representatives of the home support provider treat confidential information | at Month 6 and at Month 12
  5-point Likert scale, ranging from "completely satisfied" to "completely dissatisfied"
B.4a Specialist Physician satisfaction with the services provided by the home support provider to their patients | Month 12
  Overall satisfaction is assessed using a Visual Analog Score ranging from 0 to 10, with higher values indicating higher satisfaction.
B.4b Specialist Physician satisfaction with quantity and pertinence information provided by the home support provider on their patients | Month 12
  Satisfaction is assessed using a Visual Analog Score ranging from 0 to 10, with higher values indicating higher satisfaction.
B.5a (intervention group) Pharmacist satisfaction with the services provided by the home support provider to their patients | Month 12
  Overall satisfaction is assessed using a Visual Analog Score ranging from 0 to 10, with higher values indicating higher satisfaction.
B.5b (intervention group) Pharmacist satisfaction with the length of interactions with patients | Month 12
  Satisfaction is assessed using a Visual Analog Score ranging from 0 to 10, with higher values indicating higher satisfaction.
B.5c (intervention group) Pharmacist satisfaction with the number of interactions with patients | Month 12
  Satisfaction is assessed using a Visual Analog Score ranging from 0 to 10, with higher values indicating higher satisfaction.
B.5d (intervention group) Pharmacist perception of the usefulness of their increased role in diabetes management | Month 12
  Visual Analog Score ranging from 0 to 10, with higher values indicating higher levels of perceived usefulness.
C.1 Self-reported ability to use their insulin delivery system(pump or closed loop) [Comparison: Enhanced Care vs Standard Care] | monthly from Baseline (Month 0) to Month 12
  3 Visual Analog Scores ranging from 0 to 10s on pump or closed loop use :
  * device management
  * use of basic device functions
  * use of advanced device functions Higher scores indicate better ability to use the device.
Physician assessment of patient's ability to use their insulin delivery system (pump or closed loop [Comparison: Enhanced Care vs Standard Care] | Month 12
  3 Visual Analog Scores on physician's assessment of the patient's ability to use their insulin delivery system:
  * device management
  * use of basic device functions
  * use of advanced device functions Higher scores indicate better perceived ability to use the device.
C.3a Patient satisfaction with treatment as measured by the Diabetes Treatment Satisfaction Questionnaire - status (DTSQs) [Comparison: Enhanced Care vs Standard Care] | Baseline (Month 0) and at Month 12
  The Diabetes Treatment Satisfaction Questionnaire status (DTSQs) is an 8-question tool widely used in routine practice. Higher scores indicate higher satisfaction with their treatment.
C.3b Patient perception of treatment burden [Comparison: Enhanced Care vs Standard Care] | Baseline (Month 0) and at Month 12
  The Timkl-1 questionnaire is a 9-question tool used to assess patients' treatment burden, need for an enhanced care service, and quality of life.
  This outcome uses the treatment burden subscore, for which higher scores indicate a greater burden.
D.1 Time in the glycemic target range [Comparison: Enhanced Care vs Standard Care] | Month 12
  Time in the glycemic target range (Time-in-range or TIR) is an intuitive metric that denotes the amount of time in percentage that a person's glucose level remains within the proposed target range.
  Using measurements from continuous or flash glucose monitoring systems, TIR is the percentage of data points between 70 and 180 mg/dL.
  Complementary metrics are used:
  * Time below range (TBR) = percentage of data points < 54 mg/dL
  * Time above range (TAR) = percentage of data points > 180 mg/dL
Percentage of glycated hemoglobin (HbA1c) [Comparison: Enhanced Care vs Standard Care] | at Baseline (Month 0) and at Month 12
  The HbA1c test is used to evaluate a person's level of glucose control. The test shows an average of the blood sugar level over the past 90 days and represents a percentage. Higher values tend to indicate worse levels of glucose control.
E.1 Patient quality of life [Comparison: Enhanced Care vs Standard Care] | at Baseline (Month 0) and at Month 12
  The Timkl-1 questionnaire is a 9-question tool used to assess patients' treatment burden, need for an enhanced care service, and quality of life.
  This outcome uses the quality of life subscore, for which higher scores indicate a better quality of life.
E.2 Number and relevance of impact that can have an impact on diabetes [Comparison: Enhanced Care vs Standard Care] | monthly between Baseline (Month 0) and Month 12
  * (intervention group) Number and relevance of clinical or non-clinical events reported by the patient to the pharmacist
  * Number and relevance of clinical or non-clinical events reported by patients to their specialist doctor
  * Number and relevance of clinical or non-clinical events reported by the patient (ePRO)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno GUERCI, MD PhD, Principal Investigator — CHU NANCY; Gérard REACH, MD PhD, Study Chair — Université Sorbonne Paris Nord
Locations (1):
- CHU Nice - Hôpital l'Archet 2, Nice, Paca, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: study portal — https://prodiab1.sanoia.com/